CLINICAL TRIAL: NCT00992680
Title: A Prospective, Randomized, Multicenter, Open Label, Pilot Study to Evaluate the ROX Anastomotic Coupler System in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Pilot Study to Evaluate the ROX Anastomotic Coupler System in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: US-01
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Disease; Chronic Airflow Obstruction; Chronic Bronchitis; Pulmonary Emphysema; Walk
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Bronchitis, Chronic; Pulmonary Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Anastomotic Coupler System + standard of care per GOLD
  Interventions: Device: ROX Anastomotic Coupler System (ACS)
- Group B (No Intervention): Standard of care per GOLD alone

INTERVENTIONS:
Device: ROX Anastomotic Coupler System (ACS) — The ACS will be used to create an arteriovenous fistula in the iliac region (between the iliac artery and vein)
  Arms: Group A

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary performance of the ROX Anastomotic Coupler System (ACS), with standard of care (as defined per GOLD) in patients with Chronic Obstructive Pulmonary Disease (COPD) as compared to standard of care alone.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic disease that leads to irreversible changes in the lung structure, but also to systemic changes in the body that can influence the severity of the disease. The irreversible changes to the lungs can be seen in limitations to the pulmonary function. The purpose of this clinical investigation is to evaluate the performance and efficacy of the ROX percutaneous Anastomotic Coupler System.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Chronic Obstructive Pulmonary Disease (COPD) must be made on the basis of current findings, medical history and physical examination.

Exclusion Criteria:

* Subjects not meeting Stage III or IV Chronic Obstructive Pulmonary Disease (COPD)
* Subjects with significant comorbidities
* Subjects not qualifying because of physical or psychological condition that may put them at risk of participating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improvement in exercise capacity. | 3mo, 6mo, and 12mo

SECONDARY OUTCOMES:
Incidence of complications and adverse events. | 3mo, 6mo, and 12mo

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Pulmonary Associates, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Orlando Regional Health Care System, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Veritas Clinical Specialties, LTD, Topeka, Kansas
  - Franklin Square Hospital, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oklahoma State University Medical Center, Tulsa, Oklahoma

REFERENCES:
- [Background] Cooper CB, Celli B. Venous admixture in COPD: pathophysiology and therapeutic approaches. COPD. 2008 Dec;5(6):376-81. doi: 10.1080/15412550802522783. PMID 19353352
- [Derived] Faul J, Schoors D, Brouwers S, Scott B, Jerrentrup A, Galvin J, Luitjens S, Dolan E. Creation of an iliac arteriovenous shunt lowers blood pressure in chronic obstructive pulmonary disease patients with hypertension. J Vasc Surg. 2014 Apr;59(4):1078-83. doi: 10.1016/j.jvs.2013.10.069. Epub 2014 Jan 28. PMID 24484754